CLINICAL TRIAL: NCT00293462
Title: Management of Mucositis With GM-CSF (Sargramostim) Mouthwash Study Protocol
Brief Title: GM-CSF Mouthwash for Preventing and Treating Mucositis in Patients Undergoing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marilyn Dodd (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Marilyn Dodd, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000459510; UCSF-H452-26184-03 (Other: University of California, San Francisco); 02802 (Other: University of California, San Francisco); 5R01CA107080 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Head and Neck Cancer; Mucositis Oral; Radiation Toxicity; Tongue Cancer
Keywords: Recurrent squamous, basal cell carcinoma of the pharynx,larynx,lip; Oropharynx, paranasal sinus and nasal cavity; Stage I-IV lymphoepithelioma of the nasopharynx; Stage I-IV lymphoepithelioma of the oropharynx; Recurrent esthesioneuroblastoma of paranasal sinus, nasal cavity; Recurrent inverted papilloma of the paranasal sinus, nasal cavity; Recurrent midline granuloma of the paranasal sinus, nasal cavity; Untreated, current, metastatic squamous neck cancer; Recurrent verrucous carcinoma of the larynx; Recurrent lymphoepithelioma of the oropharynx; Stage I verrucous carcinoma of the larynx; Recurrent verrucous carcinoma of the oral cavity; Stage I verrucous carcinoma of the oral cavity; Stage II verrucous carcinoma of the larynx; Stage II verrucous carcinoma of the oral cavity; Stage III verrucous carcinoma of the larynx; Stage III verrucous carcinoma of the oral cavity; Stage IV verrucous carcinoma of the larynx; Stage IV verrucous carcinoma of the oral cavity; Recurrent adenoid cystic carcinoma of the oral cavity; Stage I adenoid cystic carcinoma of the oral cavity; Stage II adenoid cystic carcinoma of the oral cavity; Stage III adenoid cystic carcinoma of the oral cavity; Stage IV adenoid cystic carcinoma of the oral cavity; Recurrent mucoepidermoid carcinoma of the oral cavity; Stage I mucoepidermoid carcinoma of the oral cavity; Stage II mucoepidermoid carcinoma of the oral cavity; Stage III mucoepidermoid carcinoma of the oral cavity; Stage IV mucoepidermoid carcinoma of the oral cavity; Recurrent squamous cell carcinoma of the lip and oral cavity; Stage I squamous cell carcinoma of the lip and oral cavity; Stage II squamous cell carcinoma of the lip and oral cavity; Stage III squamous cell carcinoma of the lip and oral cavity; Stage IV squamous cell carcinoma of the lip and oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis; Radiation Injuries; Tongue Neoplasms; Esthesioneuroblastoma, Olfactory | interventions — sargramostim; Salts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I: GM-CSF Group (GG) (Active Comparator): Arm I: Patients were randomized to receive oral sargramostim (GM-CSF) mouthwash as a prevention, holding it in their mouths and swallowing it in intervals over 1 hour once daily. If they develop mucositis, they continue receiving GM-CSF treatment continues during 6-7 weeks of radiotherapy and until the mucositis heals.
  Interventions: Biological: sargramostim
- Arm II: Salt & Soda Group (SS) (Active Comparator): Arm II: Patients were randomized to receive salt and soda (SS) mouthwash as a prevention, holding it in their mouths and swallowing it in intervals over 1 hour once daily. If they develop mucositis, they continue receiving SS treatment continues during 6-7 weeks of radiotherapy and until the mucositis heals.
  Interventions: Other: oral salt and soda mouthwash
- Arm III: Salt & Soda Switched to GM-CSF (SG) (Active Comparator): Arm III: Patients were randomized to receive oral salt and soda (SS) mouthwash as a prevention, holding it in their mouths and swallowing it in intervals over 1 hour once daily. If they develop mucositis, they continue receiving GM-CSF treatment continues during 6-7 weeks of radiotherapy and until the mucositis heals.
  Interventions: Biological: sargramostim; Other: oral salt and soda mouthwash

INTERVENTIONS:
Biological: sargramostim
  Arms: Arm I: GM-CSF Group (GG); Arm III: Salt & Soda Switched to GM-CSF (SG)
Other: oral salt and soda mouthwash — Patients receive oral salt and soda mouthwash, holding it and swallowing it in intervals over 1 hour once daily.
  Arms: Arm II: Salt & Soda Group (SS); Arm III: Salt & Soda Switched to GM-CSF (SG)

SUMMARY:
GM-CSF may protect normal cells from the side effects, such as mucositis, of radiation therapy and may help damaged tissue heal faster after radiation therapy. This randomized clinical trial is studying how well GM-CSF works in preventing and treating mucositis in patients who are undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of radiotherapy (RT)-induced oral mucositis of any grade, using the Radiation Therapy Oncology Group Acute Radiation Morbidity Scoring Criteria (RTOG ARMSC)-Mucous Membrane, in patients treated with 1 of 2 mouthwashes (sargramostim [GM-CSF] or salt and soda). (prevention portion of the study)
* Compare the effectiveness of the 2 mouthwashes in treating oral mucositis as defined by the incidence of RTOG ARMSC-Mucous Membrane grade 3 and 4 mucositis in patients in 1 of 3 groups (salt and soda, continuing GM-CSF, or new GM-CSF). (treatment portion of the study)

Secondary

* Compare the effectiveness of the 2 mouthwashes in preventing RT-induced oral mucositis by the following direct indices:

  * Cumulative RT dose prior to onset of oral mucositis (prevention portion only)
  * Severity of RT-induced oral mucositis at onset and during treatment (using Oral Mucositis Assessment Scale (OMAS))
  * Severity of oral mucositis-related pain at onset and during treatment (using OMAS)
  * Incidence of oral mucositis-related infection at onset and during treatment (using OMAS)
  * Severity of oral mucositis-related problems with ingestion of food and fluids at onset and during treatment (using OMAS)
  * Time to healing of RT-induced oral mucositis.
* Evaluate patients using the following indirect indices of oral mucositis morbidity during the prevention and treatment portions of the study.

  * Tolerance to RT regimen
  * Functional status
  * Quality of life.

OUTLINE: This is a multicenter, randomized, controlled, double-blinded study. Patients are stratified according to radiotherapy dose schedule (standard vs hyperfractionation vs intensity modulation) and concurrent chemotherapy (yes vs no).

* Prevention (no mucositis): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral sargramostim (GM-CSF) mouthwash, holding it in their mouths and swallowing it in intervals over 1 hour once daily.
  * Arm II: Patients receive oral salt and soda mouthwash, holding it and swallowing it in intervals over 1 hour once daily.

Treatment in both arms continues during 6-7 weeks of radiotherapy and/or the onset of mucositis. Patients also perform PRO-SELF: Mouth Aware (PSMA) twice daily.

* Treatment (onset of mucositis): Patients who are currently using GM-CSF mouthwash continue use as in prevention. Patients who are currently using salt and soda mouthwash are randomized to 1 of 2 treatment arms.

  * Arm III: Patients receive GM-CSF mouthwash as in arm I.
  * Arm IV: Patients receive salt and soda mouthwash as in arm II. In both arms, treatment continues until the mucositis heals. Patients perform PSMA four times daily during and for 3 months after radiotherapy.

Quality of life is assessed at baseline and periodically after radiotherapy.

After completion of study treatment, patients are followed every once a month for 3 months.

ELIGIBILITY:
Inclusion Criteria

* Histopathologically confirmed diagnosis of head and neck cancer
* Scheduled to undergo continuous course of conventional or hyperfractionated radiotherapy or intensity-modulated radiotherapy (IMRT) with or without concurrent chemotherapy
* Planning to receive a total radiation dose ≥ 5,500 centigray (cGy), administered in a single daily fraction of 180-220 cGy (5 days a week) or twice daily fractions of 110-150 cGy
* Normal baseline oral examinations (no pre-existing lesion)
* Karnofsky performance status 60-100%
* Mentally capable of participating in research protocol
* Expected survival > 4.5 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* Aspartate aminotransferase (AST) < 5 times upper limit of normal
* HIV negative

Exclusion Criteria

* No unresolved adverse event from previous therapy
* No prior radiotherapy to the head and neck
* No prior or concurrent brachytherapy
* No prior participation in this study
* No T1 or T2 glottic tumors
* No other serious concurrent medical illness
* No history of insulin-dependent diabetes mellitus
* No prior hypersensitivity reaction to yeast material
* No recent history of oral ulceration, herpes simplex, oral candidiasis, severe gingivitis, active or chronic mucositis, or xerostomia
* No current New York Heart Association class II-IV congestive heart failure
* Not pregnant or nursing
* No chemotherapy, radiotherapy, or other investigational drugs within the past 4 weeks
* No major surgery within the past 2 weeks
* No systemic sargramostim (GM-CSF) within the past 7 days
* No systemic filgrastim (G-CSF) within the past 24 hours
* No systemic long-acting pegfilgrastim within the past 14 days
* No antibiotics, antifungals, or antivirals for oral conditions at baseline
* No other concurrent chemotherapy agent
* No concurrent enrollment on other head and neck studies
* No other concurrent investigational drugs
* No concurrent administration of any of the following:

  * "Magic or miracle mouthwash" containing a palliative mixture of topical anesthetics/analgesics, coating agents, and other medications without an approved indication for topical oral use except liquid antacid formulations (e.g., Maalox® or Mylanta® or their generic equivalents)
  * Other concurrent over-the-counter or prescription mouthwashes beyond the systematic oral care protocol provided by the study or any other drugs or agents to aid in oral hygiene (e.g., chlorhexidine, gluconate, pilocarpine, amifostine, sucralfate tablets or slurry, or benzydamine)
  * Use of corticosteroids for chronic conditions OR within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-06-07 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylin J. Dodd, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult (> 18 years of age) with confirmed histopathological diagnosis of head and neck carcinoma were recruited at the University of California, San Francisco Radiation Oncology Clinic, the Helen Diller Comprehensive Cancer Center, Saint Francis Medical Center in San Francisco, and Temple University Radiation Oncology Clinic in Philadelphia from May 2005 to Dec 2009.
Pre-assignment Details: Of 532 potential subjects that were screened, 374 were excluded as they did not meet the inclusion criteria, 45 refused to participate and 22 were no-shows (declined radiation therapy), thereby reducing our original target sample population to 91.
Period: Overall Study
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
Started | 31 | 29 | 31
Completed | 24 | 21 | 19
Not Completed | 7 | 8 | 12
Not completed — Withdrawal by Subject | 4 | 3 | 8
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Change Treatment Regimen (ineligible) | 1 | 0 | 0
Not completed — Hypersensitive Reaction (to Salt & Soda) | 0 | 1 | 0
Not completed — Refuse Radiation Treatment | 1 | 0 | 0
Not completed — No Show | 0 | 0 | 1
Not completed — Went back to his home country | 0 | 0 | 1
Not completed — Blood clot after chemotherapy | 0 | 0 | 1
Not completed — Ischemic stroke after chemotherapy | 0 | 0 | 1
Not completed — Possible Tracheostomy leakage | 0 | 1 | 0
Not completed — Low radiation dose in oral cavity | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: GM-CSF Group (GG): Arm I: Patients receive oral sargramostim (GM-CSF) mouthwash, holding it in their mouths and swallowing it in intervals over 1 hour once daily. Treatment continues during 6-7 weeks of radiotherapy and until the mucositis heals.
- Arm II: Salt & Soda Group (SS): Arm II: Patients receive oral salt and soda mouthwash, holding it and swallowing it in intervals over 1 hour once daily. Treatment continues during 6-7 weeks of radiotherapy and until the mucositis heals.
- Arm III: Salt & Soda Switched to GM-CSF (SG): Arm II patients are split, with Arm III being switched to GM-CSF when they develop mucositis.
- Total: Total of all reporting groups
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG) | Total
Number analyzed (Participants) | 31 | 29 | 31 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 26 | 77
  >=65 years | 6 | 3 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.55 (13.73) | 54.69 (12.22) | 56.26 (11.29) | 54.48 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 11 | 24
  Male | 20 | 27 | 20 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 30 | 28 | 27 | 85
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 6 | 5 | 21
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 2 | 4 | 0 | 6
  White | 18 | 16 | 22 | 56
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Number of Participants With Grade 1 or 2 Oral Mucositis (GM-CSF and SS Groups Only)
Description: The number of participants with recorded grade 1 (mild; Irritation, may experience slight pain, not requiring analgesic) or grade 2 (moderate; Patchy mucositis that may produce inflammatory serosanguinitis discharge; may experience moderate pain requiring analgesia) oral mucositis using the Radiation Therapy Oncology Group (RTOG) Acute Radiation Morbidity Scoring Criteria Oral Mucosa Assessment Scale at baseline and during radiotherapy will be recorded. The RTOG grading is reliant on a clinician's ability to judge the anatomical changes associated with oral mucositis (size and characteristics of ulceration), with symptoms ranging from Grade 0 (no symptoms) to Grade 4 (Ulceration, hemorrhage, or necrosis). A comparison of incidence in the GM-CSF Group (GG) and Arm II: Salt & Soda Group (SS) will be reported.
Time Frame: From baseline to onset of mucositis, approximately 16 days
Population: Intent to treat population consisted of randomized subjects who completed baseline questionnaire and had at least one dose of mouthwash
Measure: Number; unit: participants
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS)
Number analyzed (Participants) | 28 | 53
participants | 28 | 46
Statistical Analysis 1: Comparison: Arm I: GM-CSF Group (GG) vs Arm II: Salt & Soda Group (SS); Fisher's exact two tailed test; Test type: Superiority or Other; p = 0.09, Fisher Exact; Two by two table was used. One cell had expected frequency test less than five, so Fisher's exact two-tailed test was used

2. Primary Outcome: Comparison of the Mean Number of Days for Mucositis to Heal Across by Group
Description: The mean number of days for mucositis to heal will be used to evaluate the effectiveness of the two mouthwashes in treating oral mucositis as defined by the incidence of Radiation Therapy Oncology Group Acute Radiation Morbidity Scoring.
Time Frame: From onset of mucositis to healing of mucositis, approximately 80 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
Number analyzed (Participants) | 28 | 21 | 19
days | 81.5 (63.43) | 79.4 (31.24) | 77.4 (37.40)
Statistical Analysis 1: Comparison: Arm I: GM-CSF Group (GG) vs Arm II: Salt & Soda Group (SS) vs Arm III: Salt & Soda Switched to GM-CSF (SG); Kaplan-Meier estimate of the survival curves used information from subjects who develop mucositis to the healing of the mucositis in three groups, Group GG, SS, and SG. In order to compare the three curves that were created, the Mantel-Haenszel log-rank statistic was used; Test type: Superiority or Other; p = 0.92, Mantel Haenszel; Log rank, Breslow, Tarone-Ware test, but used mantel cox log rank for this analysis

3. Secondary Outcome: Comparison of the Combined Mean Score on the Overall Quality of Life Questionnaires by Group
Description: Quality of life at baseline, during radiotherapy, and once a month for 3 months after radiotherapy. The items on the quality of life questionnaire developed for the study range in scores from 0-10 with higher scores indicating a better quality of life. Scores at all time points were combined to compute one mean score for overall quality of life during the study.
Time Frame: Up to 3 months
Population: Of the intent to treat population, subjects who did not fill out the baseline quality of life questionnaires were not included in our analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
Number analyzed (Participants) | 28 | 25 | 27
score on a scale | 6.91 (1.59) | 6.80 (1.46) | 6.77 (1.53)
Statistical Analysis 1: Comparison: Arm I: GM-CSF Group (GG) vs Arm II: Salt & Soda Group (SS) vs Arm III: Salt & Soda Switched to GM-CSF (SG); Multilevel regression was used; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis — 0.28 (quadratic); Restricted Maximum Likelihood Methods with random intercepts was the only model used for the three groups and seven measurement time points

4. Secondary Outcome: Comparison of Combined Mean Score on the Karnofsky Performance Status Scale (KPS) by Group
Description: Functional status of participants was measured by administering the KPS which contains items asking about performing daily activities. The scores are grouped in 10s ranging from 100 (Normal, no complaints) to 0 (Dead), with higher scores indicating better functional status. The KPS was administered at baseline, during radiotherapy, and once a month for 3 months after radiation therapy. Scores at all time points were combined to compute one mean to determine overall performance status during the course of the study.
Time Frame: Up to 3 months
Population: Of the intent to treat population, subjects who did not fill out the baseline Karnofsky functional scales were not included in our analysis. They withdrew from the study after signing the consent forms for personal reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
Number analyzed (Participants) | 28 | 25 | 26
score on a scale | 84.52 (12.61) | 82.93 (10.92) | 83.49 (12.49)
Statistical Analysis 1: Comparison: Arm I: GM-CSF Group (GG) vs Arm II: Salt & Soda Group (SS) vs Arm III: Salt & Soda Switched to GM-CSF (SG); Test type: Superiority or Other; p = 0.78, Mixed Models Analysis — 0.78 (quadratic); [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Comparison of Combined Mean Score on the Pain Questionnaire by Group
Description: Severity and quality of pain was measured using a pain questionnaire developed for this study with total scores ranging from 0 (no pain) to 10 (most intense pain) with higher scores indicating a greater level of pain. The questionnaire was administered at baseline, during radiotherapy, and once a month for 3 months after radiotherapy. Scores at all time points were combined to compute one mean to determine overall pain intensity score during the course of the study
Time Frame: Up to 3 months
Population: Of the intent to treat population, subjects who did not fill out the baseline pain questionnaires were not included in our analysis. They withdrew from the study after signing the consent forms for personal reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
Number analyzed (Participants) | 27 | 25 | 27
score on a scale | 2.15 (2.40) | 1.72 (2.26) | 2.15 (2.65)
Statistical Analysis 1: Comparison: Arm I: GM-CSF Group (GG) vs Arm II: Salt & Soda Group (SS) vs Arm III: Salt & Soda Switched to GM-CSF (SG); Test type: Superiority or Other; p = 0.22, Mixed Models Analysis — 0.22 (quadratic); [statistical method as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: Serious Adverse Events and adverse events were collected in the safety population which is comprised of all participants who were both randomized and received at least one dose of the study medication. Number of participants at risk represents the number of participants who received study medications.
Arm/Group | Arm I: GM-CSF Group (GG) | Arm II: Salt & Soda Group (SS) | Arm III: Salt & Soda Switched to GM-CSF (SG)
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/28 | 2/28
Other Adverse Events (participants affected / at risk) | 18/29 | 26/28 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: GM-CSF Group (GG) (N=29) | Arm II: Salt & Soda Group (SS) (N=28) | Arm III: Salt & Soda Switched to GM-CSF (SG) (N=28)
Other (General disorders) | 0 (0) | 0 (0) | 1 (1) — Other (withdrawal symptoms-opioid)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mucositis Oral:Hypersensitivity Reaction from Salt and Soda Mouthwash
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Reactive oral mucositis : Due to the timing of the adverse event (AE), the study team determined that the reactive oral mucositis is unlikely to be related to radiation therapy and was part of the salt and soda group.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: GM-CSF Group (GG) (N=29) | Arm II: Salt & Soda Group (SS) (N=28) | Arm III: Salt & Soda Switched to GM-CSF (SG) (N=28)
Transfusion (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Sinus tachycardia due to Acetaminophen-codeine medication.
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — (Shoulder and neck area)
Other (General disorders) | 0 (0) | 0 (0) | 1 (1) — (Withdraweal symptoms-opioid)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — (Right foot)
Sinusitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — (left parotid gland)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — (bicycle accident)
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (4)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) — (>15 lbs; more than 10%)
Dehydration (Metabolism and nutrition disorders) | 5 (16) | 13 (27) | 10 (21) — (hydrated at doctor's office during/after radiation treatment)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Had the potential to have bone growth and had previous history. Based on physician's decision. Patient was in Salt and Soda group. This was not related to the mouth wash medication.
Ischemia Cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — (chest congestion)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngopharyngeal Dyesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — (mucous)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — (Asymptomatic; clinical observations only; intervention not indicated; tracheostomy area)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — (due to fentanyl patch)
Rash acne form (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — (lung biopsy)
Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) — (Percutaneous endoscopic gastrostomy tube insertion)
Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — (PEG tube removal)
Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — (basal cell carcinoma remove from thumb)
Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — (facial reconstruction)
Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — (Septoplasty)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No